CLINICAL TRIAL: NCT00666653
Title: Effects of a Dopamine Agonist on Pharmacodynamics of Levodopa in Parkinson's Disease: a Double-Blind Placebo Controlled Crossover Study
Brief Title: Effects of a Dopamine Agonist on Pharmacodynamics of Levodopa in Parkinson's Disease
Acronym: DALI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Matthew Brodsky M.D., Oregon Health & Science University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 697
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Last update posted 2008-04-25 (Estimated); Status verified 2008-04

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Dopamine Agonist; Levodopa; Pharmacokinetics; Dyskinesia
MeSH Terms: conditions — Parkinson Disease; Dyskinesias | interventions — Pramipexole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: pramipexole

SUMMARY:
The purpose of this study is to determine whether there is a benefit to giving a dopamine agonist to a patient with Parkinson's disease who is already being treated with levodopa.

DETAILED DESCRIPTION:
Patients with idiopathic PD based on London Brain Bank criteria as determined by an OHSU movement disorder specialist entered the study. They gave informed consent to a protocol approved by the Oregon Health and Science University Institutional Review Board and General Clinical Research Center (GCRC) Review Committee.

Patients were on long-term levodopa therapy, and had motor fluctuations and dyskinesia as determined during screening. Subjects were screened with finger tapping (FT) in the practically defined OFF motor state, having been off LD overnight, and in the practically defined ON motor state. To qualify, they had to have a minimum 10% improvement in the ON state.

The trial was a randomized, double-blind, placebo-controlled crossover study with subjects on pramipexole for 4 weeks and an identically appearing placebo for 4 weeks. The response to two-hour LD infusions at 0.5 (threshold) and 1.0 (suprathreshold) mg/kg/hr were examined at the end of each 4 week treatment period.

The primary outcome was finger-tapping speed, as a surrogate marker of bradykinesia, over a seven hour time period. The area under the curve (AUC) was calculated as finger taps x minutes (FTM). Secondary outcomes measured included peak motor response, as measured by FT, walking speed, dyskinesia, time-to-ON (defined as a 10% increase in finger tapping speed over the baseline), and effects of LD infusion on subjects' perceived mood, anxiety and fatigue.

Subjects were randomized to receive either pramipexole (PPX) or placebo for the initial 5 weeks of the study. The PPX and placebo was titrated up over 9 days to a target dose of 1.0mg TID. If they were already taking a DA, this was tapered and discontinued while the study medication was titrated upward. Their LD was continued according to the subjects normal schedule during this time period, as well as any other antiparkinsonian medications they were taking.

After a maintenance phase of 4 weeks on study medication (PPX 1.0mg TID or placebo TID) subjects were admitted in the evening to the inpatient GCRC at OHSU. Their last LD dose was given no later than 10 pm and all other PD medications were withheld after 10 pm. They practiced FT sessions on the night of admission. At 7 AM the next morning, a dose of the study drug was given and an IV line was placed. An IV levodopa infusion was administered starting at 9 am, continuously over 2 hours at a rate of either 0.5mg/kg/hr or 1.0 mg/kg/hr. The infusion rate was blinded and randomized. The infusion was stopped at 11 am. After 2:00 PM and when subjects were deemed "off", the usual antiparkinson medications were reinstituted.

FT, tremor, walking (timed and # of steps), dyskinesia, and a "global" PD scale were measured by research nurses, and subjects completed visual analogue scales (VASs) for anxiety, fatigue and mood every 30 minutes from 7:00 AM until 2:00 PM.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-80
* Idiopathic PD Hoehn & Yahr stage 2-4,
* diagnosed by 2 of the 3 cardinal motor features
* Fluctuation response to levodopa
* Dyskinesia
* No other historical, laboratory or physical signs to suggest an alternate diagnosis
* No significant dementia, MMSE>24
* On oral levodopa therapy

Exclusion Criteria:

* dementia
* psychosis
* severe anxiety
* unstable cardiovascular disease
* uncontrolled hypertension
* history of cardiac arrhythmias
* active peptic ulcer disease
* anemia (HCT<32%)

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2003-07; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve of motor function based on finger tapping scores | 2 months

SECONDARY OUTCOMES:
Dyskinesia rating score | 2 months
Gait performance | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Matthew A Brodsky, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Derived] Brodsky MA, Park BS, Nutt JG. Effects of a dopamine agonist on the pharmacodynamics of levodopa in Parkinson disease. Arch Neurol. 2010 Jan;67(1):27-32. doi: 10.1001/archneurol.2009.287. PMID 20065126